CLINICAL TRIAL: NCT03041454
Title: A Randomized Trial to Compare the Effects of a Novel Versus Traditional Systematic Review Format on the Ability of Health Care Managers and Policy Makers to Understand and Apply Evidence
Brief Title: Testing New Formats for the Presentation of Research Evidence to Health Care Managers and Policy Makers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SMH-312381
Record Dates: First submitted 2017-01-05; First posted 2017-02-02 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Uptake of Systematic Review Evidence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel systematic review format (Experimental): A 2-page summary of systematic review content that has been designed in collaboration with policy makers and health care managers. Participants receiving the intervention will be asked to read and answer questions using a novel systematic review format.
  Interventions: Other: Novel systematic review format
- Traditional systematic review format (No Intervention): Control participants will be asked to read and answer questions using a traditional systematic review format.

INTERVENTIONS:
Other: Novel systematic review format — A 2-page summary of systematic review content that has been designed in collaboration with policy makers and health care managers.
  Arms: Novel systematic review format

SUMMARY:
The purpose of this project is to identify and use our knowledge on the barriers and facilitators to using systematic reviews (SR) by health care managers (HCM) and policy markers (PM) to develop and test a novel format for presentation of SR for HCM and PM. We will invite HCM and PM from hospitals and regional authorities in Ontario, Alberta, and British Columbia to participate in a randomized-control trial. Participants will receive a link to an online consent survey, and then be randomly allocated to receive access to a novel SR or its traditional presentation. There is no time limit to completing the task, and participants are able to save their responses and finish later. Participants are able to withdraw from the study by not completing the task.

DETAILED DESCRIPTION:
Despite advances in the conduct and reporting of traditional systematic reviews, current evidence suggests that they are used infrequently by health care managers and policy makers in decision making. Managers and policy makers have suggested that concise presentation positively affects the use of systematic reviews. The purpose of this randomized controlled trial is to assess the impact of a traditional systematic review format compared with the innovative format on the ability of health care managers and policy makers to understand the evidence in the review and apply it to a relevant health care decision making scenario.

The two end-user groups have different formatting needs and we will therefore run 2 parallel studies, randomizing each group separately. Once participants have consented to participate, a computer generated randomization process will allocate them to one of 2 arms (1:1 ratio). Participants will either receive either a traditional format or a novel format. Unequal block randomization will be used and allocation will be concealed through central assignment. Outcomes assessors will be blinded and participants will be blinded to the citation of the review so that the traditional version will not be easily accessible in its original format from the relevant journal.

This study will be the first study to engage health care managers and policy makers in the testing of formats for presentation of research evidence relevant to their needs. The results of the project will help increase the uptake of systematic review results in health care management policy decision-making, ultimately leading to informed decision making and positively impacting the health of Canadians.

ELIGIBILITY:
Inclusion Criteria:

* Health care managers from the Alberta SCNs, CAHO in Ontario, the RHAs and AQESSS in Quebec and RHAs from BC will be invited to participate.
* Policy makers/analysts from the Ontario, BC, Alberta and Quebec Ministries of Health

Exclusion Criteria:

* Health care managers or policy makers who are unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants (health care managers or policy makers) who appropriately consider and apply the evidence from each systematic review format | This measure will be assessed at the particular time the intervention is administered (i.e., at the time the participant reads the systematic review format, an average of 2 hours).
  The proportion of participants (health care managers or policy makers) who appropriately consider and apply the evidence from each systematic review format to the scenario as measured by agreement with an expert panel's recommendation. A panel of 4 health care managers or policy makers from our research team and 2 content experts. Their answers will provide the definition of appropriate application of the evidence. Two investigators who will be blind to allocation will independently determine if the participant's answer agrees with that from the expert panel. Disagreements will be resolved by a third investigator, independently. Agreement between investigators will be reported using the kappa statistic.

SECONDARY OUTCOMES:
Comprehension of the review | This measures will be assessed at the particular time the intervention is administered (i.e., at the time the participant reads the systematic review format, an average of 2 hours).
  Comprehension of the review - defined as the proportion of participants (health care managers or policy makers) who accurately define the bottom line from the systematic review as defined by an expert panel. A panel of 4 health care managers or policy makers from our research team and 2 content experts. Their answers will provide the definition of the bottom line from the systematic review. Two investigators who will be blind to allocation will independently determine if the participant's answer agrees with that from the expert panel. Disagreements will be resolved by a third investigator, independently. Agreement between investigators will be reported using the kappa statistic.
Intention to use evidence | This measures will be assessed at the particular time the intervention is administered (i.e., at the time the participant reads the systematic review format, an average of 2 hours).
  Intention to use evidence - collected through a 12-item likert scale survey. The survey has good face validity amongst policy makers and managers. The mean and SD of each item in the survey will be reported and we will provide a summary score of all items and convert it to a percentage.
Perceived tentativeness of research findings | This measures will be assessed at the particular time the intervention is administered (i.e., at the time the participant reads the systematic review format, an average of 2 hours).
  Perceived tentativeness of research findings - collected through a 6-item likert scale survey. This has been pre-tested to make sure that the items are intelligible to people and to achieve high levels of face validity and reliability. The mean and SD of each item in the survey will be reported and we will provide a summary score of all items and convert it to a percentage.
Provisional opinion about the intervention | This measures will be assessed at the particular time the intervention is administered (i.e., at the time the participant reads the systematic review format, an average of 2 hours).
  Provisional opinion about the intervention - collected through a 14-item likert scale survey. This has been pre-tested to make sure that the items are intelligible to people and to achieve high levels of face validity and reliability. The mean and SD of each item in the survey will be reported and we will provide a summary score of all items and convert it to a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon e Straus, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No